CLINICAL TRIAL: NCT07190144
Title: Coronary Flow Reserve Changes After Semaglutide Treatment
Status: Completed | Type: Observational
Sponsor: Ekrem Bilal Karaayvaz (Other)
Collaborators: MEDICANA (Unknown)
Responsible Party: Sponsor-Investigator, Ekrem Bilal Karaayvaz, Assistant Professor, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: IstanbulU-EBKaraayvaz-2
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: The Study Focused on the Vascular Effects of Semaglutide in Both Diabetic and Non-diabetic Patients; Obesity &Amp; Overweight
Keywords: Coronary Flow Reserve; Semaglutide; Diabetes Mellitus
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-diabetic patients: Non-diabetic patients who have planned to given semaglutide by an endocrinology specialist, mostly to give weight, were performed CFR with echocardiography before and 3 months after the treatment.
- Diabetic patients: Diabetic patients, who were planned to start semaglutide by an endocrinology specialist and were otherwise has same demographic data as non-diabetic patients, were performed CFR with echocardiography before and 3 months after the treatment

SUMMARY:
The goal of this observational study is to learn about the effects of semaglutide to coronary artery flow in diabetic and non-diabetic patients. The main question it aims to answer is:

Does semaglutide enhance coronary artery flow in diabetic and non-diabetic patients?

Participants already planned taking semaglutide by an endocrine specialist as their treatment was assessed with CFR before and 3 months after.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were planned to start semaglutide.

Exclusion Criteria:

* Ischemic heart disease
* Previous stent implantation or coronary bypass
* Heart failure
* Cardiomyopathies
* Inflammatory diseases
* Autoimmune rheumatic disease
* Chronic liver and renal insufficiency

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diabetic and non-diabetic and planned to start semaglutide has referred to cardiology clinic for the study.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who had acute coronary syndrome | From start of the study to 3 months after
  Semaglutide is known for its beneficial effects on coronary vasculature. If a patient had myocardial infarction, this patient can no longer participate in study because the CFR ultimately changes.

SECONDARY OUTCOMES:
Number of patients who can not lose weight | From start to 3 months
  Semaglutide is not only a diabetic drug but is also known for its weight loss properties. If the patient is unable to lose weight, additional information should be obtained as to why the drug is not working for this specific patient and should be removed from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicana International Istanbul Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Lincoff AM, Brown-Frandsen K, Colhoun HM, Deanfield J, Emerson SS, Esbjerg S, Hardt-Lindberg S, Hovingh GK, Kahn SE, Kushner RF, Lingvay I, Oral TK, Michelsen MM, Plutzky J, Tornoe CW, Ryan DH; SELECT Trial Investigators. Semaglutide and Cardiovascular Outcomes in Obesity without Diabetes. N Engl J Med. 2023 Dec 14;389(24):2221-2232. doi: 10.1056/NEJMoa2307563. Epub 2023 Nov 11. PMID 37952131